CLINICAL TRIAL: NCT03234660
Title: The Effects of Dexmedetomidine on the Neurotoxicity From General Anesthesia Assessed by Plasma Glial Fibrillary Acidic Protein
Brief Title: Dexmedetomidine and Neuroprotection in Children Undergoing General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: H1706-132-861
Record Dates: First submitted 2017-07-17; First posted 2017-07-31 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Dexmedetomidine
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine (Experimental): dexmedetomidine infusion
  Interventions: Drug: Dexmedetomidine Hydrochloride
- control (Placebo Comparator): placebo infusion
  Interventions: Other: control

INTERVENTIONS:
Drug: Dexmedetomidine Hydrochloride — dexmedetomidine 1mcg/kg loading and 0.5mcg/kg/hr continuous infusion during surgery
  Arms: Dexmedetomidine
Other: control — 0.9% normal saline continuous infusion
  Arms: control

SUMMARY:
Neuroapoptosis is induced by the administration of anesthetic agents to the young brain. Recent studies showed that the a2-adrenoceptor agonist, dexmedetomidine plays a trophic role during development and is neuroprotective in several settings of neuronal injury in animals. We hypothesized that neuroprotective effect of dexmedetomidine would be associated with evidence of brain injury detected by elevation of plasma concentration of glial fibrillary acid protein in children undergoing general anesthesia.

DETAILED DESCRIPTION:
GFAP measure

ELIGIBILITY:
Inclusion Criteria:

* children undergoing general anesthesia longer than 3 hours

Exclusion Criteria:

* past history of anesthesia
* cardiopulmonary bypass
* preexisting neurocognitive dysfunction
* abnormalities of liver profile (aspartate transaminase > 40 unit/L, alanine aminotransferase > 40 unit/L)

Ages: 1 Month to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-10-05 (Actual); Study Completion 2019-10-05 (Actual)

PRIMARY OUTCOMES:
Glial fibrillary acid protein | change from baseline glial fibrillary acid protein at 3 hours after the anesthetic induction
  plasma was collected at the given specific time

CONTACTS AND LOCATIONS:
Locations (1):
- SNUH, Seoul, Jongro Gu, South Korea